CLINICAL TRIAL: NCT04932330
Title: ICU-acquired Weakness in Extracorporeal Membrane Oxygenation Support: Frequency and Risk Factors
Brief Title: Risk Factors of ICU-acquired Weakness
Acronym: ICU-AW
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-0041
Record Dates: First submitted 2021-06-01; First posted 2021-06-21 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: ICU Acquired Weakness
Keywords: ICU Acquired Weakness; Extracorporeal Membrane Oxygenation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ICU-acquired weakness group: Patients receiving extracorporeal membrane oxygenation support who had a Medical Research Council (MRC) sum score < 48 out of a maximal score of 60 when discharged.
- no ICU-acquired weakness group: Patients receiving extracorporeal membrane oxygenation support who had a Medical Research Council (MRC) sum score ≥ 48 out of a maximal score of 60 when discharged.

SUMMARY:
We conducted a retrospective study of critical ill patients who used ECMO during their ICU stay. ICU-AW was diagnosed at the time when patients discharged and had a Medical Research Council (MRC) sum score < 48 out of a maximal score of 60. We divided patients to ICU-acquired weakness group and no ICU-acquired weakness group and compared their clinical characteristics. Baseline characteristics and therapy details were collected from the case report forms and inspection reports. Univariable analysis and logistic regression analysis were used to analyze clinical characteristics of individuals and to find risk factors of ICU-AW.

ELIGIBILITY:
Inclusion Criteria:

* Critical ill patients who used extracorporeal membrane oxygenation during their ICU stay. Patients were recruited from the general ICU of the second affiliated hospital of Zhejiang University, between March 2017 to March 2020.

Exclusion Criteria:

* Patients who was less than 18 years old, had been proven or suspected neurological impairment, using extracorporeal membrane oxygenation less than 24 hours, severe head or spinal cord injury and pregnant woman.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: There were 85 patients used extracorporeal membrane oxygenationbetween March 2017 to March 2020. Among the 85 patients, 22 patients presented exclusion criteria and 63 patients were included in the final analysis.
Sampling Method: Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Differences between ICU-acquired weakness in patients receiving extracorporeal membrane oxygenation support | 1 day
  We compared the clinical characteristics between ICU-acquired weakness group and no ICU-acquired weakness group by univariate analysis . Then we used logistic regression analysis and found out differences of ICU-acquired weakness.

SECONDARY OUTCOMES:
Frequency of ICU-acquired weakness in in patients receiving extracorporeal membrane oxygenation support | 1 day
  We calculated the prevalence of ICU-acquired weakness on the patients included in our research.

CONTACTS AND LOCATIONS:
Locations (1):
- Xinyi Chen, Hangzhou, Please Select, China

IPD SHARING:
Plan to Share IPD: Yes
One year after the article was published, and the opening lasted for one year